CLINICAL TRIAL: NCT04155359
Title: Establishment of the Performance of the miR Sentinel™ BCa Test in Men and Women Presenting for Initial Diagnosis of Bladder Cancer and the miR Sentinel™ BCR Test to Identify Recurrent Bladder Cancer
Brief Title: Clinical Evaluation of the miR Sentinel BCa™ Test to Diagnose Bladder Cancer in Hematuria Patients
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: miR Scientific LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: MIR-B001
Record Dates: First submitted 2019-11-05; First posted 2019-11-07 (Actual); Last update posted 2023-10-25 (Actual); Status verified 2023-10

CONDITIONS: Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Urine for Sentinel™ BCa Test
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of the study is to establish the clinical performance and utility of the miR Sentinel™ BCa Test, a urine exosome-based diagnostic test, as an aid in diagnosing bladder cancer. Male and female participants presenting with micro- or macro-hematuria who are undergoing cystoscopy for diagnosis of bladder cancer will be eligible for the study. Urine samples will be collected at the time of the first presentation, and the miR Sentinel™ BCa Score determined and compared to the results of cystoscopy. Participants with no evidence of cancer following cystoscopy will be designated cancer-free, while those participants with a positive cystoscopy and histopathological evidence of cancer will be designated as having bladder cancer. Participants with a positive cystoscopy who subsequently undergo TURBT will be eligible to continue in the study. Urine samples will be collected at each follow up visit for up to three years, and the miR Sentinal™ BCR Score will be determined and compared to the results of surveillance cystoscopy.

DETAILED DESCRIPTION:
Primary Objective(s):

Establish the performance characteristics of the miR Sentinel™ BCa Test as an aid in diagnosing bladder cancer in men and women presenting with hematuria.

Secondary Objective(s) Establish the performance characteristics of the miR Sentinel™ BCR Test in identifying bladder cancer patients with recurrent disease.

Study Design:

Participants who present with evidence of hematuria (micro- or macro-hematuria) and are scheduled to have cystoscopy will be enrolled. All participants will provide a urine sample for the miR Sentinel™ BCa Test prior to cystoscopy for bladder cancer. The presence or absence of cancer will be determined by cystoscopy. Diagnosis of bladder cancer will be confirmed by histopathology. The performance of the miR Sentinel™ BCa Test for classifying future patients as either bladder cancer or no bladder cancer will be established. The sensitivity, specificity, positive and negative predictive value determined for the miR Sentinel™ BCa Test and will be compared to cystoscopy.

Statistical Analysis:

Definitions. The general notation P(A | B) means the probability (prevalence) of the event A among the subgroup of patients in a population all of whom have the event B.

1. Sensitivity = P(screening test + | disease).
2. Specificity = P(screening test - | no disease).
3. PPV = P(disease | screening test + ).
4. NPV = P(no disease | screening test -).

Estimate of Sample Size. This study is targeted to enroll 3000 participants, 1500 males and 1500 females, who present with hematuria. Approximately 15% of participants with hematuria have bladder cancer; men have a higher incidence of bladder cancer than women. Therefore, the investigators anticipate that 225 males (15% of all males enrolled) and 175 females (approximately 12% of all women enrolled) will have bladder cancer confirmed by histopathology.

Overview. As outlined below, this clinical study will enroll male and female participants that have been identified as having (micro- or macro-) hematuria and are therefore at risk for bladder cancer and meet clear eligibility criteria. The study will evaluate the miR Sentinel™ BCa Test for classification of participants as cancer or no cancer, to be used as an aid in diagnosing bladder cancer. For participants diagnosed with bladder cancer who undergo TURBT will be eligible to continue in the study of miR Sentinel™ BCR Test to monitor for recurrent disease in conjunction with the cystoscopy associated with the standard of care recommended by the AUA.

The miR Sentinel™ BCa Test functions by controlling sensitivity at or above a pre-specified level, denoted 1-α; where α is the false-negative rate of the test (a patient who truly has bladder cancer has a negative test result), For example, the value that has been assumed in this design is α≤0.05 so that sensitivity is at least 95%. To describe how the cutoff for the miR Sentinel™ BCa Test is calculated to control sensitivity, for each participant determined to have bladder cancer by histopathology, the miR Sentinel™ BCa Score will be calculated using an approach that blinds each participant's true cancer status, mimicking the setting for classification of a future patient. The cutoff value for the Sentinel™ Score is then chosen so that the empirical sensitivity, calculated over all patients in the training dataset, yields a 95% upper confidence interval with lower limit 1-α.

To provide some detail on the calculation of the error rates of the test, the method to be used for estimation is cross-validation. Cross-validation produces unbiased estimators of error rates for classification of a future patient, with unknown true disease status, as the number of patients in the training dataset grows large. If there are 3000 participants with hematuria divided equally from male and female population in the study and 225 males and 175 females with bladder cancer, then, for males, the upper 95% confidence interval based on an observed empirical sensitivity of 97% (218/225) will have a lower bound of 0.95, and for females, the upper 95% confidence interval based on an observed empirical sensitivity of 98% (171/175) will have a lower bound of 0.95.

Validation of the miR Sentinel™ BCR for identifying patients with recurrent disease uses essentially the same statistical methodology. However, the classification is based on the comparison of the miR Sentinel™ BCR signature for patients with stable (non-recurrent disease) and patients with evidence of progressive (recurrent) disease. The longitudinal monitoring of participants diagnosed with bladder cancer by cystoscopy may provide additional information related to anticipatory changes in the Sentinel™ signature indicative of recurrence.

ELIGIBILITY:
Inclusion Criteria:

* Males and females between the ages of 45 and 85 years of age
* Signed informed consent prior to initiation of any study-related procedures
* Minorities are included in this protocol
* Micro- or macro-hematuria

Exclusion Criteria:

* Persons incapable of providing informed consent
* Any person with a prior history of bladder cancer
* For continued enrollment in the validation of the miR SentinelMales and females between the ages of 45 and 85 years of age BCR Test, previous malignancies including bladder cancer, treatment with chemotherapeutic of immunotherapeutic agents
* Persons with an inherited cancer syndrome or a medical history suggestive of an inherited cancer syndrome

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 3000 participants (1500 males and 1500 females) will be enrolled from multi clinical site sin the U.S. and Canada. Participants will be males and females between the ages of 45 and 85 years presented with micro- or macro-hematuria, with cystoscopy as part of routine clinical workup for diagnosis of bladder cancer.
Sampling Method: Non-Probability Sample
Enrollment: 444 (Actual)
Dates: Start 2020-10-13 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
To establish the performance characteristics of the miR Scientific Sentinel™ Bladder Cancer Diagnostic Test (miR Sentinel™ BCa Test), a urine exosome-based diagnostic test, to identify bladder cancer in participants presenting with hematuria | Urine samples will be collected from participants at the time of entry and analyzed immediately for the miR Sentinel™ BCa test. Additional urine samples will be collected and analyzed at each follow-up visit up to 1 year.
  The miR Sentinel™ BCa test is an in-vitro urine exosome-based diagnostic test. The test measures up to 280 sncRNA present in urine exosomes and produces a dichotomized assessment of "-1" (no cancer) and "+1" (cancer) based on the expression profiles of the exosomal sncRNAs As outlined in detail in the statistical analysis of the description, among the 3000 participants (1500 males; 1500 females) enrolled, it is anticipated that 2600 (1275 males; 1325 females) will have a Sentinel™ BCa Score of "-1", indicative of no cancer , and 400 (225 males; 175 females) will have a Sentinel™ BCa Score of "+1", indicative of cancer. Concordance and discordance between the final Sentinel™ BCa Score and the histopathology reports of biopsy and cystoscopy results will be used to determine the sensitivity, specificity, positive and negative predictive values of the test.

SECONDARY OUTCOMES:
Validate the performance characteristics of the miR Scientific Sentinel™ Bladder Cancer Recurrence Test (miR Sentinel™ BCR Test) for the identification of recurrent disease in a longitudinal study | Urine samples will be collected from participants at entry, prior and post TURBT, given the miR Sentinel™ BCa test is "+1". Additional urine samples will be collected and analyzed at each follow-up visit, up to three years.
  The miR Sentinel™ BCR Test is an in-vitro urine exosome-based surveillance test that uses the same 280 sncRNAs a the miR Sentinel™ BCa Test, but uses a different importance weighting of individual sncRNA entities to produce a dichotomized miR Sentinel™ BCR Score of "-1" (no recurrence) and "+1" (recurrence) that predicts recurrence in participants previously diagnosed with bladder cancer following transurethral resection of bladder tumor (TURBT). Concordance and discordance between the final Sentinel™ BCR Score and the results of surveillance cystoscopy will be used to determine the sensitivity, specificity, positive and negative predictive values of the test.

CONTACTS AND LOCATIONS:
Overall Officials: Carl A Olsson, MD, Principal Investigator — Integrated Medical Professionals
Locations (1):
- Integrated Medical Professionals, Farmingdale, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided